CLINICAL TRIAL: NCT04080193
Title: Gender-sensitive Enhancement of Common Weight Loss Strategies for Overweight and Obesity: a Personalized Smartphone App
Brief Title: Gender-sensitive Enhancement of Common Weight Loss Strategies for Overweight and Obesity
Acronym: I-GENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto-Friedrich-University Bamberg (Other)
Collaborators: Department of Psychosomatic Medicine, LWL University Hospital Bochum (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71/02060305; DRKS00016623 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2019-04-25; First posted 2019-09-06 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Overweight and Obesity; Weight Loss; Gender
Keywords: Gender; Overweight; Obesity; Intervention; Smartphone-App
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The study will be a Smartphone-based interventional trial. To assess the effectiveness of the intervention weight- and eating-related behavior and cognitive and emotional responding as well as body-weight will be assessed using questionnaires and ecological momentary assessment (EMA) for one week at a pre- (T0), post- (T1) and two follow-up-assessments after six (T2) and 12 months (T3).
  Interventions: Behavioral: Smartphone-based interventional trial
- Control Group (No Intervention): Members of the control group will participate at each assessment. During the intervention phase they will receive treatment as usual.

INTERVENTIONS:
Behavioral: Smartphone-based interventional trial — According to the SIRs the 12-week intervention will contain exercises from three out of six different key modules (e.g. self-efficacy, impulsivity). The remaining modules will be implemented as mini-modules during the end of the intervention phase. The study will be designed gender-sensitive instead of gender-dichotomous. This means that treatment contents will be individualized based on gender-related SIRs and not biological sex. Participants choose between two different styles of presentation for each module and the contents can be deepened within specific exercises.
  Arms: Intervention Group

SUMMARY:
The major aim of the proposed study is to develop a gender-sensitive individually tailored add-on intervention that focusses on improving individual gender-specific SIRs (subjective illness representations) in obese or overweight individuals. We will investigate whether this will improve compliance with and long-term success of common weight loss interventions. The effectiveness of this intervention in every-day-life with regard to weight-related behavioral changes and weight loss will be evaluated within a randomized controlled setting.To enhance the applicability of the intervention in every-day-life and its dissemination we plan to develop a smart-phone-based intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Obesity class I or II with subjectively experienced weight-related impairment and a current will to lose weight.
2. Overweight (i.e. BMI between 25 and 29.9 kg/m²) with weight-related health problems and/or visceral adipose tissue and/or high psychosocial weight-related distress with a current will to lose weight.

Exclusion Criteria:

1. Obesity Class III (i.e. BMI >39.9 kg/m²).
2. Current (or within the last 12 months) involvement in a structured weight loss intervention.
3. Insulin-dependent type 1 diabetes.
4. Previous or intended bariatric surgery.
5. Current psychotherapeutic treatment of weight-related health problems.
6. Weight-enhancing drugs.
7. Drugs which promote weight-loss (e.g. anti-obesity drugs).
8. Weight-enhancing health problems which are not yet treated.
9. Cancerous disease within the last five years.
10. Current substance-use disorders, depression, psychosis, suicidal tendency or pregnancy.
11. Severe cognitive impairments.
12. Insufficient knowledge of the german language.
13. Binge-Eating Disorder or Bulimia nervosa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in Physical Activity | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to physical activity (motion sensors) will be investigated respecting gender-related differences.
Changes in Eating Behavior | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to eating behavior (DEBQ) will be investigated respecting gender-related differences.
Changes in Subjective Illness Representations | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to subjective illness representations (IPQ-R) will be investigated respecting gender-related differences.

SECONDARY OUTCOMES:
Weight Change | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to weight will be investigated as assessed by BMI.
Changes in Emotional Competence | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to subjective feeling of emotional competence (SEK-27) will be investigated respecting gender-related differences.
Changes in Impulsivity | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to impulsivity (BIS-15) will be investigated respecting gender-related differences.
Changes in Coping Strategies | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to coping strategies (Brief COPE) will be investigated respecting gender-related differences.
Changes in Weight-Related Life Quality: ORWELL-97 | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to weight-related life quality (ORWELL-97) will be investigated respecting gender-related differences.
Changes in Self-Efficacy: General-Self-Efficacy-Scale | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to self-efficacy (General-Self-Efficacy-Scale) will be investigated respecting gender-related differences.

OTHER OUTCOMES:
Changes in General Life Quality: L-1 | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to general life quality (L-1) will be investigated respecting gender-related differences.
Changes in Weight Bias Internalization | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to weight bias internalization (WBI-Scale) will be investigated respecting gender-related differences.
Changes in General Weight Bias | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to general weight bias (Fat Phobia Scale) will be investigated respecting gender-related differences.
Changes in Psychopathology | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to psychopathology (BSI-10) will be investigated respecting gender-related differences.
Changes in Self-Esteem | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to self-esteem (Rosenberg Self-Esteem Scale) will be investigated respecting gender-related differences.
Changes in Food Addiction | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to food addiction (YFAS) will be investigated respecting gender-related differences.
Media Usage | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The potential impact of media usage (OSVe-S) on the effectiveness of the intervention as well as potential changes of media usage behaviour in the course of the intervention will be investigated.
Valuation of perceived discrimination due to physical appearance | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to subjective valuation of perceived discrimination (POTS) will be investigated respecting gender-related differences.
Social Support | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The potential impact of social support (ESSI) on the effectiveness of the intervention as well as potential changes of social support behaviour in the course of the intervention will be investigated.
Impulsive Eating Behaviour | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to impulsive eating behaviour (subscale FEV) will be investigated respecting gender-related differences.
Changes in Food Related Impulsivity | The outcome will be measured at four assessments. At the beginning of the study (day 0), after finishing the app intervention (12 weeks later) and at to follow-up assessments 6 and 12 months later.
  The effectiveness of the intervention with regard to food related impulsivity (newly developed instrument FRIS) will be investigated respecting gender-related differences.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Steins-Löber, Prof. Dr., Principal Investigator — Otto-Friedrich-University Bamberg; Stephan Herpertz, Prof. Dr., Principal Investigator — Department of Psychosomatic Medicine, LWL University Hospital Bochum; Jörg Wolstein, Prof. Dr., Principal Investigator — Otto-Friedrich-University Bamberg
Locations (2):
- Germany (2):
  - Otto-Friedrich-University, Bamberg, Bavaria
  - LWL-University Hospital Department of Psychosomatic Medicine and Psychotherapy, Bochum, North Rhine-Westphalia

REFERENCES:
- [Background] Prill S, Henning C, Schroeder S, Steins-Loeber S, Wolstein J. Does Weight-Cycling Influence Illness Beliefs in Obesity? A Gender-Sensitive Approach. J Obes. 2021 Aug 21;2021:8861386. doi: 10.1155/2021/8861386. eCollection 2021. PMID 34471546
- [Background] Henning C, Schroeder S, Steins-Loeber S, Wolstein J. Gender and Emotional Representation Matter: Own Illness Beliefs and Their Relationship to Obesity. Front Nutr. 2022 Feb 8;9:799831. doi: 10.3389/fnut.2022.799831. eCollection 2022. PMID 35211498
- [Result] Pape M, Herpertz S, Schroeder S, Seiferth C, Farber T, Wolstein J, Steins-Loeber S. Food Addiction and Its Relationship to Weight- and Addiction-Related Psychological Parameters in Individuals With Overweight and Obesity. Front Psychol. 2021 Sep 21;12:736454. doi: 10.3389/fpsyg.2021.736454. eCollection 2021. PMID 34621227
- [Derived] Pape M, Herpertz S, Farber T, Seiferth C, Schoemann N, Wolstein J, Steins-Loeber S. Food Addiction in Individuals With Overweight and Obesity Undergoing a 12-Week Long Tailored mHealth Weight Loss Intervention. Eur Eat Disord Rev. 2025 Sep;33(5):931-940. doi: 10.1002/erv.3196. Epub 2025 Apr 3. PMID 40181555
- [Derived] Schoemann N, Seiferth C, Pape M, Farber T, Herpertz S, Steins-Loeber S, Wolstein J. Improving Food-Related Inhibitory Control Through an mHealth Intervention-A Secondary Outcome Analysis of an RCT. Obes Sci Pract. 2024 Dec 2;10(6):e70026. doi: 10.1002/osp4.70026. eCollection 2024 Dec. PMID 39624149
- See also: Study Homepage — http://www.i-gendo.de